CLINICAL TRIAL: NCT03049917
Title: Financial Incentives to Increase Pediatric HIV Testing
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenyatta National Hospital (Other Government); University of Nairobi (Other)
Responsible Party: Principal Investigator, Jennifer Slyker, Assistant Professor, Department of Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000599; 323-NJU-TRIAL (Other Grant/Funding Number: International AIDS Society)
Record Dates: First submitted 2017-02-03; First posted 2017-02-10 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: HIV
Keywords: financial incentive; pediatric HIV testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No incentive (No Intervention): No incentive
- KES financial incentive 1 (Experimental): Kenyan Shillings conditional cash transfer upon HIV testing
  Interventions: Behavioral: Financial incentive
- KES financial incentive 2 (Experimental): Kenyan Shillings conditional cash transfer upon HIV testing
  Interventions: Behavioral: Financial incentive
- KES financial incentive 3 (Experimental): Kenyan Shillings conditional cash transfer upon HIV testing
  Interventions: Behavioral: Financial incentive
- KES financial incentive 4 (Experimental): Kenyan Shillings conditional cash transfer upon HIV testing
  Interventions: Behavioral: Financial incentive

INTERVENTIONS:
Behavioral: Financial incentive — Conditional cash transfer upon HIV testing
  Arms: KES financial incentive 1; KES financial incentive 2; KES financial incentive 3; KES financial incentive 4

SUMMARY:
The purpose of this study is to determine whether giving small financial incentives will motivate parents to test their children for HIV.

DETAILED DESCRIPTION:
The study will be a randomized controlled trial (RCT) with 5 arms with equal allocation to each arm: no incentive, or one of 4 different levels of financial incentive. We will randomize 800 parents with children of unknown status at HIV treatment clinics in Western Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver receiving HIV care
* Parent/caregiver has one or more children <13 years old
* Child is HIV exposed (parent/caregiver report or clinic confirmation)
* Caregiver reports child's HIV status is unknown

Exclusion Criteria:

* None

  * The investigators reserve the right to exclude any potential enrollee who is deemed to be at high personal risk, or whose children are at high personal risk, of interpersonal violence, by study participation .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Slyker, PhD, Principal Investigator — University of Washington; Irene N Njugna, MBChB, Msc, Principal Investigator — University of Washington/Kenyatta National Hospital
Locations (1):
- Kisumu County Hospital, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Open to collaboration. Please contact the study PIs for requests for data sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: January 2019
Access Criteria: Contact PIs for more info

REFERENCES:
- [Background] Wagner AD, Njuguna IN, Neary J, Omondi VO, Otieno VA, Babigumira J, Maleche-Obimbo E, Wamalwa DC, John-Stewart GC, Slyker JA. Financial Incentives to Increase Uptake of Pediatric HIV Testing (FIT): study protocol for a randomised controlled trial in Kenya. BMJ Open. 2018 Oct 3;8(10):e024310. doi: 10.1136/bmjopen-2018-024310. PMID 30287676
- [Background] Njuguna IN, Wagner AD, Omondi VO, Otieno VA, Neary J, Bosire R, Babigumira JB, Levin C, Maleche-Obimbo E, Wamalwa DC, John-Stewart G, Slyker J. Financial Incentives for Pediatric HIV Testing in Kenya. Pediatr Infect Dis J. 2018 Nov;37(11):1142-1144. doi: 10.1097/INF.0000000000002035. PMID 29596217
- [Background] Atkins DL, Wagner AD, Zhang J, Njuguna IN, Neary J, Omondi VO, Otieno VA, Ondeng'e K, Wamalwa DC, John-Stewart G, Slyker JA, Beima-Sofie K. Brief Report: Use of the Consolidated Framework for Implementation Research (CFIR) to Characterize Health Care Workers' Perspectives on Financial Incentives to Increase Pediatric HIV Testing. J Acquir Immune Defic Syndr. 2020 May 1;84(1):e1-e6. doi: 10.1097/QAI.0000000000002323. PMID 32049774
- [Derived] Njuguna IN, Wagner AD, Neary J, Omondi VO, Otieno VA, Orimba A, Mugo C, Babigumira JB, Levin C, Richardson BA, Maleche-Obimbo E, Wamalwa DC, John-Stewart G, Slyker J. Financial incentives to increase pediatric HIV testing: a randomized trial. AIDS. 2021 Jan 1;35(1):125-130. doi: 10.1097/QAD.0000000000002720. PMID 33048877
- Available data/document: Study Protocol: Current FIT Protocol — https://depts.washington.edu/globalwach/wordpress/wp-content/uploads/2020/12/2.18.18-FIT-Protocol_V4.0_clean_.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- No Incentive: KES financial incentive = $0
- KES Financial Incentive 1: KES financial incentive 1= $1.25
- KES Financial Incentive 2: KES financial incentive 2= $2.50
- KES Financial Incentive 3: KES financial incentive 3= $5
- KES Financial Incentive 4: KES financial incentive 4= $10
Period: Overall Study
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4
Started | 90 | 89 | 93 | 92 | 88
Completed | 31 | 31 | 44 | 51 | 54
Not Completed | 59 | 58 | 49 | 41 | 34

BASELINE CHARACTERISTICS:
Groups:
- No Incentive: KES financial incentive= $0
- Total: Total of all reporting groups
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4 | Total
Number analyzed (Participants) | 90 | 89 | 93 | 92 | 88 | 452
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 90 | 89 | 93 | 92 | 88 | 452
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.5 [31 to 47] | 37 [30 to 45] | 38 [32 to 45] | 38 [32 to 45] | 39.5 [32 to 48] | 38 [32 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 62 | 65 | 55 | 59 | 305
  Male | 26 | 27 | 28 | 37 | 29 | 147
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 90 | 89 | 93 | 92 | 88 | 452
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Overall number of baseline participants [Count of Participants; unit: Participants] | 90 | 89 | 93 | 92 | 88 | 452

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Present Children for HIV Testing
Description: Number of caregivers who present child(ren) to complete HIV testing at the study clinic within 2 months of recruitment; test results will be recorded in a study questionnaire
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- No Incentive: KES financial incentive=$0
- KES Financial Incentive 1: KES financial incentive 1=$1.25
- KES Financial Incentive 2: KES financial incentive 2=$2.50
- KES Financial Incentive 3: KES financial incentive 3=$5
- KES Financial Incentive 4: KES financial incentive 4=$10
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4
Number analyzed (Participants) | 90 | 89 | 93 | 92 | 88
Participants | 31 | 31 | 44 | 51 | 54

2. Primary Outcome: Number of Days Participants Take to Bring Children for HIV Testing
Description: Number of days it took between randomization and caregiver presenting the child for HIV testing
Time Frame: 2 months
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- No Incentive: KES financial incentive =$0
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4
Number analyzed (Participants) | 90 | 89 | 93 | 92 | 88
days | 8 [3 to 23] | 7 [4 to 14] | 4 [1 to 11] | 5 [2 to 14] | 5 [2 to 8]

3. Secondary Outcome: Number of Female Participants Who Present Children for HIV Testing (Females)
Description: HIV testing [primary outcome 1] stratified by caregiver sex (females)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- KES Financial Incentive 1: KES financial incentive 1=$1.25 Females
- KES Financial Incentive 2: KES financial incentive 2: $2.50 Females
- KES Financial Incentive 3: KES financial incentive 3:$5 Females
- KES Financial Incentive 4: KES financial incentive 4:$10 Females
- All Females: Total females enrolled
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4 | All Females
Number analyzed (Participants) | 64 | 62 | 65 | 55 | 59 | 305
Participants | 25 | 22 | 34 | 29 | 38 | 156

4. Secondary Outcome: Number of Male Participants Who Present Children for HIV Testing
Description: Time to HIV testing [primary outcome 1] stratified by caregiver sex (males)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- KES Financial Incentive 2: KES financial incentive 2:$2.50 Females
- All Males: Total males enrolled
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4 | All Males
Number analyzed (Participants) | 26 | 27 | 28 | 37 | 29 | 147
Participants | 6 | 9 | 10 | 22 | 16 | 55

5. Secondary Outcome: Number of Caregivers With One Child Who Present Children for HIV Testing
Description: HIV testing [primary outcome 1] stratified by number of children (one child)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- KES Financial Incentive 2: KES financial incentive 2=$2.50 Females
- KES Financial Incentive 3: KES financial incentive 3=$5 Females
- KES Financial Incentive 4: KES financial incentive 1=$10
  Females
- All With One Child: Caregivers with one child
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4 | All With One Child
Number analyzed (Participants) | 42 | 41 | 33 | 36 | 38 | 190
Participants | 15 | 14 | 26 | 29 | 32 | 90

6. Secondary Outcome: Number of Participants With More Than 1 Child Who Present Children for HIV Testing
Description: Number of participants presenting children for HIV testing among caregivers with more than child
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- KES Financial Incentive 4: KES financial incentive 4=$10 Females
- All With More Than One Child: All families with more than one child
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4 | All With More Than One Child
Number analyzed (Participants) | 47 | 48 | 58 | 55 | 49 | 257
Participants | 15 | 17 | 16 | 21 | 21 | 116

7. Secondary Outcome: Number of Caregivers With Age Less Than Median Presenting Children for HIV Testing
Description: Number of participants presenting for HIV testing stratified by caregiver age (caregiver <=38 years)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- No Incentive: No incentive upon HIV testing for child
- KES Financial Incentive 1; KES Financial Incentive 2; KES Financial Incentive 3; KES Financial Incentive 4: Kenyan Shillings conditional cash transfer upon HIV testing
  Financial incentive: Conditional cash transfer upon HIV testing
  Females
- All With Caregiver Age <=38 Years: Uptake of testing if Caregiver age <=38 years
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4 | All With Caregiver Age <=38 Years
Number analyzed (Participants) | 47 | 50 | 50 | 47 | 43 | 237
Participants | 15 | 19 | 22 | 26 | 26 | 108

8. Secondary Outcome: Number of Caregivers With Age More Than Median Presenting Children for HIV Testing
Description: Number of caregivers presenting children for HIV testing stratified by caregiver age (caregiver >38 years)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- No Incentive: No incentive with uptake of child HIV testing
- All With Caregiver Age >38 Years: Uptake of testing if Caregiver age >38 years
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4 | All With Caregiver Age >38 Years
Number analyzed (Participants) | 43 | 39 | 43 | 45 | 45 | 215
Participants | 16 | 12 | 22 | 25 | 28 | 103

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | No Incentive | KES Financial Incentive 1 | KES Financial Incentive 2 | KES Financial Incentive 3 | KES Financial Incentive 4
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/89 | 0/93 | 0/92 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/89 | 0/93 | 0/92 | 0/88
Other Adverse Events (participants affected / at risk) | 0/90 | 0/89 | 0/93 | 0/92 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03049917/Prot_SAP_000.pdf